CLINICAL TRIAL: NCT03049293
Title: Measurement of Midazolam Levels in Follicular Fluid and Correlation of Midazolam Levels in Follicular Fluid and Oocyte Quality, Fertilization Rate, Embryo Development Pattern and Euploid Status
Brief Title: Measurement of Midazolam Levels in Follicular Fluid
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Difficulty in recruiting participants
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Prof Dr. Human Fatemi, Medical Director, ART Fertility Clinics LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1610-ABU-074-HF
Record Dates: First submitted 2017-01-12; First posted 2017-02-10 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Midazolam Overdose
Keywords: COPD,IVF
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group using Propofol (No Intervention): Sedation will be established by administering 100mcs of Fentanyl, and 1-1.5mg/kg of body weight of Propofol.
- Study group Midazolam group (Experimental): Sedation will be established by administering Midazolam 1mg, 100mcs of Fentanyl, and 0.5-1mg/kg of body weight of Propofol. Further boluses of Propofol will be given according to the need of the patient and time consumed for oocyte retrieval.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam — The impact of Midazolam levels in follicular fluid.
  Arms: Study group Midazolam group

SUMMARY:
To determine the impact of Midazolam levels in follicular fluid on morpho-kinetics and morpho-genetics.

The reason to measure Midazolam levels in larger size follicles in this study is to maximize the chances to get a mature oocyte and therefore develop into a potential embryo to be analyzed.

DETAILED DESCRIPTION:
The correlation of Midazolam levels in follicular fluid and euploid status of the embryos is worth exploring as no data exists that suggests any influence on the quality of the embryos from using this substance for IVF since its earliest days. Measuring time lapsed from injection to first oocyte retrieval as well as time lapsed in between first and last oocyte retrieved will grand insight into the rise of levels of Midazolam inside the follicular fluid, correlated with the chromosomal status and the morphokinetic development of the euploid embryos.

ELIGIBILITY:
Inclusion Criteria:

* Infertility (prim. / sec.)
* Age >18 - ≤ 38 years.
* BMI 19-30
* Stimulation in GnRH-antagonist protocol, using rFSH
* Expected normal ovarian response (6)
* At least 4 follicles with the size ≥ than 17 mm on the day of OPU
* Patients undergoing PGS
* Able to understand the aim of the study and to provide consent

Exclusion Criteria:

* History of endometriosis, classified according to the American Fertility Society (AFS) as stage 3 or more.
* Severe male factor

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Midazolam values measured by the time from the injection of Midazolam to the oocyte aspiration . | 6-12 months
  To determine the impact of Midazolam levels in follicular fluid on morpho-kinetics and morpho-genetics.

CONTACTS AND LOCATIONS:
Overall Officials: Human Mo Fatemi, MD, Principal Investigator — IVI Middle East Clinic
Locations (1):
- IVI Middle East Fertilty Clinic, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Follicular fluid levels of midazolam, fentanyl, and alfentanil during transvaginal oocyte retrieval. — https://www.ncbi.nlm.nih.gov/pubmed/7589618
- See also: Midazolam/ketamine sedative combination compared with fentanyl/propofol/isoflurane anaesthesia for oocyte retrieval. — https://www.ncbi.nlm.nih.gov/pubmed/10402383